CLINICAL TRIAL: NCT06096727
Title: Energize! Internet-Delivered Physical Activity Program for Adults with Knee Replacement
Brief Title: The Energize! Study for Adults with Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00130186
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthroplasty
Keywords: physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Energize! (Experimental): Participants randomized to Energize! will start the program immediately after baseline.
  Interventions: Behavioral: Energize!
- Delayed Energize! (Other): Participants randomized to Delayed Energize! will start the program after the 3 month assessment.
  Interventions: Behavioral: Energize!

INTERVENTIONS:
Behavioral: Energize! — Energize! is 3 month online physical activity program which consists of weekly physical activity goals, video lessons, action planning, and homework.

SUMMARY:
The purpose is to examine the effects of an online physical activity program on moderate to vigorous intensity physical activity, pain, and physical function in adults with knee replacement at 3 months (post-intervention) and 6 months (maintenance).

DETAILED DESCRIPTION:
Participants with knee replacement will be randomized to start the online physical activity program (Energize!) either immediately or after 3 months. The online program consists of weekly physical activity goals, video lessons, action planning, and homework to help increase physical activity to 200 min/week. Assessments will be completed at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have had a partial or total knee replacement ≥12 months ago
* Have regular access to the internet
* Willing to wear activity monitor for 7 days at baseline, 3 & 6 months
* Engage in less than 60 minutes of self-reported moderate intensity exercise

Exclusion Criteria:

* Have a mobility limiting comorbidity
* Non-English speaking
* Have a scheduled surgery within the next 6 months that would limit activity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate to vigorous intensity physical activity | baseline to 3 months
  activity assessed by Actigraph accelerometers
Pain intensity | baseline to 3 months
  Pain intensity assessed by Patient-Reported Outcomes Measurement Information System pain intensity survey. 0 represents no pain and 10 reports the most severe pain
Self-reported physical function | baseline to 3 months
  Physical function assessed by Patient-Reported Outcomes Measurement Information System physical function/mobility survey. A t-score of 0 represents poor function compared to average and 100 represents better function.

SECONDARY OUTCOMES:
Minutes of moderate to vigorous intensity physical activity | 3 months to 6 months
  activity assessed by Actigraph accelerometers
Pain intensity | 3 months to 6 months
  Pain intensity assessed by Patient-Reported Outcomes Measurement Information System pain intensity survey. 0 represents no pain and 10 reports the most severe pain
Self-reported physical function | 3 months to 6 months
  Physical function assessed by Patient-Reported Outcomes Measurement Information System physical function/mobility survey. A t-score of 0 represents poor function compared to average and 100 represents better function.

OTHER OUTCOMES:
Adherence to Energize program - video lessons viewed | 3 months
  Number of video lessons viewed
Adherence to Energize program - planning or reporting exercise minutes | 3 months
  Number of weeks exercise minutes were planned or reported
Adherence to Energize program - homework assignments | 3 months
  Number of homework assignments completed

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, we do not have a plan to share IPD.